CLINICAL TRIAL: NCT05131594
Title: Immune Response to Post Acute Sequelae of SARSCoV2: a Correlation of Clinical Symptoms and Inflammatory Pathways
Brief Title: Evaluating the Response of the Immune System of People with Long COVID (post SARS-CoV-2)
Acronym: LCRC
Status: Enrolling by invitation | Type: Observational
Sponsor: Huntington Memorial Hospital (Other)
Collaborators: San Diego Biomedical Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00054801
Record Dates: First submitted 2021-11-19; First posted 2021-11-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: COVID-19
Keywords: post-acute sequelae of SARS-CoV2; post-acute COVID-19 syndrome; long COVID
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Many people who have had COVID 19 continue to experience symptoms long after they have recovered from the acute infection. This study will examine the clinical symptoms of people with "Long COVID" and measure various markers of inflammation in their blood.

DETAILED DESCRIPTION:
Patients who attend the Long Covid Recovery Clinic at Huntington Hospital will be offered participation in the study. After giving written informed consent, their medical history along with a description of clinical symptoms given through an extensive questionnaire will be accessed. Venous blood will be collected as a baseline and then at follow up visits (as dictated by changes in clinical symptomatology) for evaluation of corollary immune parameters. Patients will be followed at a minimum of every 2 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in Huntington Hospital's Long Covid Recovery Clinic
* Documented previous infection with SARS-CoV2
* Symptoms suggestive of post-acute sequelae of SARS-CoV2 (including but not limited to chronic fatigue, brain fog, muscle and joint pain, cardiac and pulmonary issues, or other factors related to their acute COVID-19 event)
* Signed Informed Consent Form

Exclusion Criteria:

* No documented positive SARS-CoV2 serologies
* No post-acute sequelae of SARS-CoV2 symptomatology
* Incarcerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (18 years old or older) who enroll in Huntington Hospital's Long Covid Recovery Clinic will be offered but are under no obligation to participate in this study. Subjects will have documented previous infection with SARS-CoV2 and symptoms suggestive of post-acute sequelae of SARS-CoV2 (including but not limited to chronic fatigue, brain fog, muscle and joint pain, cardiac and pulmonary issues, or other factors related to their acute COVID-19 event).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-10-13 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Correlation of symptomatology with inflammatory profiles in patients with Post-Acute Sequelae of SARS-CoV2 (PASC) | From onset of infection to 24 months
  Do patient symptoms correlate with abnormalities in inflammatory profiles?
Identification of immunologic and inflammatory features of PASC based on results of immunologic and inflammatory assays | From onset of infection to 24 months
  Are there abnormalities in immunologic and inflammatory assays unique to PASC?
Evaluation and delineation of the pathologic pathways and long-term effects of SARS-CoV2 infection | From onset of infection to 60 months
  What are the pathological pathways and long-term effects of SARS-CoV2?
Identification of risks factor for PASC | From onset of infection to 24 months
  What are the risk factors for PASC?
Identification of potential sites of therapeutic intervention to ameliorate symptomatology of PASC | From onset of infection to 60 months
  Are there potential sites of therapeutic intervention to relieve the symptoms of PASC?

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Shriner, MD, Principal Investigator — Huntington Hospital
Locations (1):
- Huntington Hospital, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: No